CLINICAL TRIAL: NCT03665181
Title: Crystalline Exposition During Pediatric Cranial CT Imaging
Acronym: ECTOPIC
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Commission of the French Radiology (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2018/11
Record Dates: First submitted 2018-09-07; First posted 2018-09-11 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Any Pathology Requiring a Cranial CT Imaging
Keywords: Radioprotection; dosimetry; tomodensitometry; pediatrics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- without modification of dose and without bismuth mask: The cranial CT imaging presrcibed in usual care will be performed without modification of dose and without bismuth mask
  Interventions: Other: use or non-use of dose modulator and bismuth mask
- with modification of dose and with bismuth mask: e cranial CT imaging presrcibed in usual care will be performed with modification of dose and with bismuth mask
  Interventions: Other: use or non-use of dose modulator and bismuth mask
- without modification of dose and with bismuth mask: e cranial CT imaging presrcibed in usual care will be performed without modification of dose and with bismuth mask
  Interventions: Other: use or non-use of dose modulator and bismuth mask
- with modification of dose and without bismuth mask: e cranial CT imaging presrcibed in usual care will be performed with modification of dose and without bismuth mask
  Interventions: Other: use or non-use of dose modulator and bismuth mask

INTERVENTIONS:
Other: use or non-use of dose modulator and bismuth mask — For each child for who the eligibility criteria are met, the CT exam is perfomed with or without dose modulator associated to with or without bismuth mask

SUMMARY:
This study focuses on reduction of X-rays dose applied to eye's lens during cranial CT in children. Principal objective is to analyse the efficiency of ocular bismuth masks, which are associated with an eye's lens dose modulation

DETAILED DESCRIPTION:
Eye's lens radiosensitivity represents an important subject of investigation in radiology. Indeed, eye's lens is recognised as one of the most radiosensitive organs in human body.[1,2] Radiation induced cataracts represent a determining effect of ionising radiations and has been widely studied. "International Commission for Radiological Protection" has evaluated cataract appearance threshold at 15 Gy in 1977 ",[3] then at 8 Gy [4] and 5 Gy in 2007.[5] Finally, in 2011 new studies gave rise to a new limit of appearance of 0.5 Gy. Eye's lens radiosensitivity seems to have been underestimated for several years and so there is a significant improvement to be made in radioprotection in order to protect to the best of the investigator's ability both patient and manipulator. This was also confirmed by the Directive EURATOM 2013/59 (which is in the process of being transposed in French legislation)[6] that reduces legal limit dose delivered to eye's lens from 150mSv to20mSv, for categories A workers.

This study is performed on 4 sequential groups, of ten patients, whereby one control group without ocular protection added. Other groups benefit either from a bismuth ocular protection, from a dose modulation applied to the eye's lens, or from both techniques associated. For each group, experiment is then focused on dose received by the eye's lens (measured using TLD detectors) as well as on Image quality obtained. Currently, there is no recommendation regarding lens protection for patient who benefit of a head tomodensitometry. Some practices are already used routinely but without a critical analysis of a comparison of their respective benefits.

ELIGIBILITY:
Inclusion Criteria:

* Children between 5 and 16 yrs old
* Indication of cerebral CT with or without contrast regardless to indication or exam specificity
* Patients beneficiary or affiliated to health system security
* Oral consent for data processing from the child and his/her representative of parental authority

Exclusion Criteria:

* Children anxious or agitated
* Sedated patients or patients under general anaesthesia
* Impossibility to position the skull on the orbito-meatal plane (intubation for example)
* Patients under legal protection

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The population include all children for who a cranial CT imaging will be required within usual care in the radiology ward of Bordeaux University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2020-10-27 (Actual)

PRIMARY OUTCOMES:
Efficiency of a bismuth based ocular protection associated with eye's lens dose modulation technique | Baseline
  quantification of the efficiency of a bismuth based ocular protection associated with eye's lens dose modulation technique during cranial CT of children. This will be measured by the average dose difference relative to the number of helices, kV and mAs delivered between groups 1 and 2

SECONDARY OUTCOMES:
Efficiency of a bismuth based ocular protection | Baseline
  Quantification of the efficiency of a bismuth based ocular protection during CT acquisition. This will be measured by the average dose difference relative to the number of helices, kV and mAs delivered between groups 1 and 3
Efficiency of eye's lens dose modification | Baseline
  Quantification of the efficiency of eye's lens dose modification technique during CT acquisition. This will be measured by the average dose difference relative to the number of helices, kV and mAs delivered between groups 1 and 4
Image quality | Baseline
  Quantitative analysis of the image quality obtained with both systems after CT acquisition. Quality will be assessed by radiologist's categorization

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No